CLINICAL TRIAL: NCT01808339
Title: A Randomised, Repeat-dose, Placebo-controlled, Three-way Crossover, Double Dummy Study to Evaluate and Compare the Efficacy of Fluticasone Furoate Inhalation Powder Delivered Via the Single Strip Dry Powder Inhaler When Administered Either in the Morning or in the Evening, in Male and Female Asthmatic Subjects
Brief Title: To Investigate the Effects of Altering the Time of Day of Dosing (Morning or Evening) With Fluticasone Furoate 100 Micrograms Once Daily Administered Via a Dry Powder Inhaler in Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 117156
Record Dates: First submitted 2013-02-21; First posted 2013-03-11 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Fluticasone Furoate, FF Inhalation Powder, morning dosing, evening dosing, efficacy, FEV1
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FF AM dose (Experimental): All the subjects in this study will take part in 3 treatment periods and will receive all three treatments (one per period) in a random manner. In one of the treatment periods, subjects will receive FF 100 mcg in the morning (approximately 09:00) and placebo in the evening (approximately 21:00) for 14 days (+/- 2 days).
  Interventions: Drug: Fluticasone Furoate (FF); Drug: Placebo
- FF PM dose (Experimental): All the subjects in this study will take part in 3 treatment periods and will receive all three treatments (one per period) in a random manner. In one of the treatment periods, subjects will receive FF 100 mcg in the evening (approximately 21:00) and placebo in the morning (approximately 09:00) for 14 days (+/-2 days).
  Interventions: Drug: Fluticasone Furoate (FF); Drug: Placebo
- Placebo (Placebo Comparator): All the subjects in this study will take part in 3 treatment periods and will receive all three treatments (one per period) in a random manner. In one of the treatment periods, subjects in this arm will receive Placebo in the evening and morning (at approximately 09:00 and 21:00) for 14 days (+/- 2 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone Furoate (FF) — Inhalation powder 100 microgram per blister strip to be administered via dry powder inhaler either in the morning (AM dose with FF and PM dose with +/-2 days).
  Arms: FF AM dose; FF PM dose
Drug: Placebo — Placebo in single strip to be administered via dry powder inhaler in the morning and evening for 14 days (+/- 2 days).

SUMMARY:
This study will investigate the effects of altering the time of day of dosing (morning or evening) with Fluticasone Furoate 100 (FF 100) micrograms (mcg) once daily administered via a dry powder inhaler (DPI) in subjects with persistent bronchial asthma. This is a repeat-dose, double-blind, randomized, placebo-controlled, three-way crossover study to compare the effect of morning (AM) and evening (PM) dosing with FF 100 on lung function. Twenty-four male and female subjects with persistent bronchial asthma will be enrolled to ensure twenty evaluable subjects. The three treatments will be FF 100 AM (with placebo PM), FF 100 PM (with placebo AM) and matching placebo (AM and PM). All treatments will be administered for 14 (+/-2) days with 14 day run-in and 14 to 21 day washout periods. The total duration of the study will be approximately 13 to18 weeks for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a documented history of persistent asthma, with the exclusion of other significant pulmonary diseases (pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma).
* Male or female between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is:
* Of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy or postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use contraception method, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotropin (hCG) test at screening and serum or urine hCG test prior to dosing and agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until completion of the follow up visit or has only same-sex partners, when this is her preferred and usual lifestyle.
* All subjects must either be clinically stable on a low to mid dose inhaled corticosteroid (ICS) (with or without a short acting beta-2 receptor agonist [SABA]) such as Fluticasone Propionate (FP) 100 to250 mcg twice-daily (total daily dose 200 to 500 mcg) or equivalent, for at least 4 weeks preceding the screening visit or be clinically stable on a low dose ICS/ long acting beta-2 receptor agonist (LABA) combination, such as SERETIDE/ADVAIR 100/50 twice- daily or equivalent (administered either in combination or from separate inhalers), for at least 4 weeks preceding the screening visit. Higher ICS/LABA doses (i.e. equivalent to SERETIDE/ADVAIR 250/50 or 500/50) would not be acceptable. Subjects must refrain from using their LABA for at least 24 hour (h) prior to the screening visit
* Subjects with a screening pre-bronchodilator FEV1 >= 60 percent of predicted. Predicted values will be based upon National Health and Nutrition Examination Survey (NHANES III).
* During the screening visit, subjects must demonstrate the presence of reversible airway disease, defined as an increase in FEV1 of >= 12.0 percent over baseline and an absolute change of >= 200 mL within 60 minutes following 4 inhalations of albuterol/salbutamol inhalation aerosol (or equivalent nebulized treatment with albuterol/salbutamol solution).
* All subjects must be able to replace all their current asthma treatments with albuterol/salbutamol aerosol inhaler at screening for use as needed for the run-in period and throughout the duration of the study. Subjects on LABAs must also withhold this for at least 24 h prior to the screening visit. Subjects will therefore be on SABA alone for the duration of the study, and on SABA and FF during the FF treatment periods. Subjects must be able to withhold albuterol/salbutamol for at least 6 h prior to screening and study visits.
* Subjects who are current non-smokers and who have a pack history of <= 10 pack years. A subject may not have used inhaled tobacco products within the past 3 months (i.e., cigarettes, cigars or pipe tobacco).
* Body weight >= 50 kilograms (kg) and Body Mass Index (BMI) within the range 19.0 to29.9 kg/meter^2 (inclusive)
* Based on single or averaged QT duration corrected for heart rate by Fridericia's formula (QTcF) values of triplicate electrocardiograms (ECGs) obtained over a brief recording period: QTcF < 450 millisecond (msec); or QTcF < 480 msec in subjects with Bundle Branch Block.
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2x Upper limit of normal (ULN), alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Able to satisfactorily use the DPI

Inclusion Criteria for Randomisation to Treatment

* Evening pre-dose FEV1 of >=60 percent of their predicted normal at Day 1
* Daily diary compliance defined as completion of all AM daily diary data on >=4 of the last 7 consecutive days of the Run-in Period (not including the date of randomisation) and completion of all PM daily diary data on >=4 of the last 7 consecutive days of the Run-in Period (not including the date of randomisation)

Exclusion Criteria:

* A history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 5 years.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of screening and led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Any asthma exacerbation requiring oral corticosteroids within 12 weeks of screening or that resulted in overnight hospitalization requiring additional treatment for asthma within 6 months prior to screening.
* A subject has any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study. The list of additional excluded conditions/diseases includes, but is not limited to the following: congestive heart failure, known aortic aneurysm, clinically significant coronary heart disease, clinically significant cardiac arrhythmia, stroke within 3 months of Visit 1, uncontrolled hypertension, recent or poorly controlled peptic ulcer, hematologic, hepatic, or renal disease (with the exception of Gilbert's syndrome or asymptomatic gallstones), immunologic compromise, current malignancy, tuberculosis (current or untreated), Cushing's disease, Addison's disease, uncontrolled diabetes mellitus, uncontrolled thyroid disorder, recent history of drug or alcohol abuse.
* Any adverse reaction including immediate or delayed hypersensitivity to any beta 2 agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the DPI (i.e. lactose).
* History of severe milk protein allergy.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Subjects who have taken oral steroids within 12 weeks of the screening visit.
* History of regular alcohol consumption within 6 months of the study defined as Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a 285 mL glass of full strength beer or 425 mL schooner of light beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine.

Exclusion Criteria based upon diagnostic assessments

* A subject will not be eligible if he/she has clinical visual evidence of oral candidiasis at screening.
* Pregnant females as determined by positive serum hCG test at screening or by positive serum or urine hCG test prior to dosing.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody. Other Criteria
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product (IP) within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* No subject is permitted to perform night shift work for 1 week prior to screening until completion of the study treatment periods.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Exclusion Criteria for Randomisation to Treatment

* Resuming their asthma medication (excluding albuterol/salbutamol inhalation aerosol provided at screening).
* Occurrence of a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear during the run-in period that led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Evidence of a severe exacerbation, defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension or injection) for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids between screening and Day 1.
* Clinical visual evidence of oral candidiasis at Day 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kempsford RD, Bal J, Baines A, Renaux J, Ravindranath R, Thomas PS. The efficacy of fluticasone furoate administered in the morning or evening is comparable in patients with persistent asthma. Respir Med. 2016 Mar;112:18-24. doi: 10.1016/j.rmed.2015.12.011. Epub 2016 Jan 12. PMID 26823210
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 117156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants meeting eligibility criteria at the Screening visit entered a 2-week Run-in Period for Baseline safety evaluations and to obtain measures of asthma status.
Pre-assignment Details: Participants meeting randomization criteria were enrolled in the study for 13-18 weeks: three 14-day treatment periods separated by a 14- to 21-day washout period, followed by a follow-up visit within 7-14 days of the last dose.
Groups:
- FF 100 µg AM /FF 100 µg PM/Placebo: Participants received 3 treatments (A, B, and C) in sequence ABC. During treatment A participants received fluticasone furoate (FF) 100 micrograms (100 µg) in the morning (AM) at approximately 09:00 and received placebo in the evening (PM) at approximately 21:00 for 14 days (+/-2 days) via a dry powder inhaler (DPI). During treatment B participants received placebo in the AM and FF 100 µg in the PM for 14 days (+/-2 days) via a DPI. During treatment C participants received placebo via a DPI for 14 days (+/-2 days) in the AM and PM. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FF 100 µg AM/Placebo/FF 100 µg PM: Participants received 3 treatments (A, B, and C) in sequence ACB. During treatment A participants received FF 100 µg in the AM at approximately 09:00 and received placebo in the PM at approximately 21:00 for 14 days (+/-2 days) via a DPI. During treatment B participants received placebo in the AM and FF 100 µg in the PM for 14 days (+/-2 days) via a DPI. During treatment C participants received placebo via a DPI for 14 days (+/-2 days) in the AM and PM. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FF 100 µg PM /FF 100 µg AM/Placebo: Participants received 3 treatments (A, B, and C) in sequence BAC. During treatment A participants received FF 100 µg in the AM at approximately 09:00 and received placebo in the PM at approximately 21:00 for 14 days (+/-2 days) via a DPI. During treatment B participants received placebo in the AM and FF 100 µg in the PM for 14 days (+/-2 days) via a DPI. During treatment C participants received placebo via a DPI for 14 days (+/-2 days) in the AM and PM. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FF 100 µg PM /Placebo/FF 100 µg AM: Participants received 3 treatments (A, B, and C) in sequence BCA. During treatment A participants received FF 100 µg in the AM at approximately 09:00 and received placebo in the PM at approximately 21:00 for 14 days (+/-2 days) via a DPI. During treatment B participants received placebo in the AM and FF 100 µg in the PM for 14 days (+/-2 days) via a DPI. During treatment C participants received placebo via a DPI for 14 days (+/-2 days) in the AM and PM. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- Placebo/FF 100 µg AM/FF 100 µg PM: Participants received 3 treatments (A, B, and C) in sequence CAB. During treatment A participants received FF 100 µg in the AM at approximately 09:00 and received placebo in the PM at approximately 21:00 for 14 days (+/-2 days) via a DPI. During treatment B participants received placebo in the AM and FF 100 µg in the PM for 14 days (+/-2 days) via a DPI. During treatment C participants received placebo via a DPI for 14 days (+/-2 days) in the AM and PM. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- Placebo/FF 100 µg PM /FF 100 µg AM: Participants received 3 treatments (A, B, and C) in sequence CBA. During treatment A participants received FF 100 µg in the AM at approximately 09:00 and received placebo in the PM at approximately 21:00 for 14 days (+/-2 days) via a DPI. During treatment B participants received placebo in the AM and FF 100 µg in the PM for 14 days (+/-2 days) via a DPI. During treatment C participants received placebo via a DPI for 14 days (+/-2 days) in the AM and PM. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
Period: Treatment Period 1 (14 Days)
Arm/Group | FF 100 µg AM /FF 100 µg PM/Placebo | FF 100 µg AM/Placebo/FF 100 µg PM | FF 100 µg PM /FF 100 µg AM/Placebo | FF 100 µg PM /Placebo/FF 100 µg AM | Placebo/FF 100 µg AM/FF 100 µg PM | Placebo/FF 100 µg PM /FF 100 µg AM
Started | 4 | 4 | 4 | 4 | 6 | 6
Completed | 4 | 3 | 4 | 2 | 4 | 5
Not Completed | 0 | 1 | 0 | 2 | 2 | 1
Not completed — Met Protocol-defined Stopping Criteria | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0
Period: Washout Period 1 (14-21 Days)
Arm/Group | FF 100 µg AM /FF 100 µg PM/Placebo | FF 100 µg AM/Placebo/FF 100 µg PM | FF 100 µg PM /FF 100 µg AM/Placebo | FF 100 µg PM /Placebo/FF 100 µg AM | Placebo/FF 100 µg AM/FF 100 µg PM | Placebo/FF 100 µg PM /FF 100 µg AM
Started | 4 | 3 | 4 | 2 | 4 | 5
Completed | 4 | 3 | 4 | 2 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (14 Days)
Arm/Group | FF 100 µg AM /FF 100 µg PM/Placebo | FF 100 µg AM/Placebo/FF 100 µg PM | FF 100 µg PM /FF 100 µg AM/Placebo | FF 100 µg PM /Placebo/FF 100 µg AM | Placebo/FF 100 µg AM/FF 100 µg PM | Placebo/FF 100 µg PM /FF 100 µg AM
Started | 4 | 3 | 4 | 2 | 4 | 5
Completed | 4 | 3 | 4 | 2 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (14-21 Days)
Arm/Group | FF 100 µg AM /FF 100 µg PM/Placebo | FF 100 µg AM/Placebo/FF 100 µg PM | FF 100 µg PM /FF 100 µg AM/Placebo | FF 100 µg PM /Placebo/FF 100 µg AM | Placebo/FF 100 µg AM/FF 100 µg PM | Placebo/FF 100 µg PM /FF 100 µg AM
Started | 4 | 3 | 4 | 2 | 4 | 5
Completed | 4 | 3 | 4 | 2 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (14 Days)
Arm/Group | FF 100 µg AM /FF 100 µg PM/Placebo | FF 100 µg AM/Placebo/FF 100 µg PM | FF 100 µg PM /FF 100 µg AM/Placebo | FF 100 µg PM /Placebo/FF 100 µg AM | Placebo/FF 100 µg AM/FF 100 µg PM | Placebo/FF 100 µg PM /FF 100 µg AM
Started | 4 | 3 | 4 | 2 | 4 | 5
Completed | 4 | 3 | 3 | 2 | 4 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Met Protocol-defined Stopping Criteria | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FF 100 µg AM/FF 100 µg PM/Placebo: Participants received 3 treatments (A, B, and C) in either of the six sequences: ABC , ACB, BAC, BCA, CAB, or CBA. During treatment A participants received fluticasone furoate (FF) 100 micrograms (100 µg) in the morning (AM) at approximately 09:00 and received placebo in the evening (PM) at approximately 21:00 for 14 days (+/-2 days) via a dry powder inhaler (DPI), during treatment B: participants received placebo in the AM and FF 100 µg in the PM for 14 days (+/-2 days) via a DPI during treatment C: participants received placebo via a DPI for 14 days (+/-2 days) in the AM and PM. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
Arm/Group | FF 100 µg AM/FF 100 µg PM/Placebo
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (10.99)
Gender [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1
  Asian - Central/South Asian Heritage | 2
  Asian - South East Asian Heritage | 1
  White - White/Caucasian/European Heritage | 21
  White - Mixed Race | 1
  Mixed Race | 2

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean Forced Expiratory Volume in 1 Second (FEV1) Measured Over 24 Hours at Day 14 of Each Treatment Period
Description: FEV1 is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured using site equipment (KoKo Pneumotach Spirometer). Weighted mean FEV1 was calculated using the Day 14 24-hour serial FEV1 measurements taken at 3, 6, 9, 12, 15, 18, 21, and 24 hours post-dose (measured in the evening of Day 15). At each time point, the highest of three technically acceptable measurements was recorded. FEV1 weighted mean was analyzed using a mixed effects analysis of a covariance model with fixed effect terms for treatment and period, participant Baseline, period Baseline, gender, and age as covariates, and participant as a random effect.
Time Frame: 24 hours post-PM dose on Day 14 of each treatment period (up to Study Day 105)
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study medication, and had at least one Baseline and post-dose FEV1 measurement performed. Only those participants with non-missing covariates and a post-Baseline FEV1 measurement were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- FF 100 µg AM: Participants received fluticasone furoate (FF) 100 micrograms (100 µg) in the morning (AM) at approximately 09:00 and received placebo in the evening (PM) at approximately 21:00 for 14 days (+/-2 days) via a dry powder inhaler (DPI) in one of the three treatment periods. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FF 100 µg PM: Participants received placebo in the AM at approximately 09:00 and FF 100 µg in the PM at approximately 21:00 for 14 days (+/-2 days) via a DPI in one of the three treatment periods. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- Placebo: Participants received placebo via a DPI for 14 days (+/-2 days) in the AM and PM. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
Arm/Group | FF 100 µg AM | FF 100 µg PM | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Liters | 3.303 (0.0589) | 3.332 (0.0584) | 3.227 (0.0585)
Statistical Analysis 1: Comparison: FF 100 µg AM vs Placebo; Test type: Superiority or Other; Median Difference (Final Values) = 0.077, 90% CI 2-sided [0.001 to 0.152] — The estimated value represents the difference in Least Squares Means between FF 100 µg AM and Placebo (FF 100 µg AM minus Placebo)
Statistical Analysis 2: Comparison: FF 100 µg PM vs Placebo; Test type: Superiority or Other; Median Difference (Final Values) = 0.105, 90% CI 2-sided [0.029 to 0.180] — The estimated value represents the difference in Least Squares Means between FF 100 µg PM and Placebo (FF 100 µg PM minus Placebo)
Statistical Analysis 3: Comparison: FF 100 µg AM vs FF 100 µg PM; Test type: Superiority or Other; Median Difference (Final Values) = -0.028, 90% CI 2-sided [-0.102 to 0.045] — The estimated value represents the difference in Least Squares Means between FF 100 µg AM and FF 100 µg PM (FF 100 µg AM minus FF 100 µg PM)

2. Secondary Outcome: Pre-treatment AM and PM Trough FEV1 on Day 14 of Each Treatment Period
Description: FEV1 is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured using site equipment (KoKo Pneumotach Spirometer). FEV1 PM trough FEV1 values were the values taken pre-treatment on Day 14, and AM trough FEV1 values were the values taken pre-treatment on Day 15 in each treatment period; thus, there is only one value (pre-treatment record) per period for AM and PM trough.
Time Frame: Day 14 of each treatment period (up to Study Day 105)
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study medication, and had at least one Baseline and post-dose FEV1 measurement performed. Only those participants available at the specified time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF 100 µg AM | FF 100 µg PM | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Liters
  AM Trough FEV1 | 3.299 (0.0707) | 3.359 (0.0702) | 3.286 (0.0703)
  PM Trough FEV1 | 3.236 (0.0607) | 3.290 (0.0598) | 3.177 (0.0600)

3. Secondary Outcome: Number of Participants With Any Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs were collected from the start of dosing with investigational product and until follow-up.
Time Frame: Up to 18 weeks
Population: All Subjects Population: all participants who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | FF 100 µg AM | FF 100 µg PM | Placebo
Number analyzed (Participants) | 23 | 24 | 25
Participants | 18 | 18 | 16

4. Secondary Outcome: Peak Expiratory Flow (PEF)
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. AM and PM pre-treatment PEF was measured throughout the study for the purposes of monitoring participants' asthma stability, and was measured from the start of the Run-in Period until completion of Treatment Period 3 (including during the washout periods), prior to study medication and/or any rescue albuterol/salbutamol inhalation aerosol use. The data collected were only assessed by the Investigator on an individual basis during the study and were not formally summarized or statistically analyzed; consequently, data are not reported.
Time Frame: Up to 18 weeks
Arm/Group | FF 100 µg AM | FF 100 µg PM | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse event (SAE) and non serious AEs were collected from the start of dosing with investigational product until follow-up (up to 18 weeks).
Description: SAEs and non-serious AEs are reported for the Safety Population, comprised of all participants randomized to treatment, who had taken at least one dose of study medication.
Arm/Group | FF 100 µg AM | FF 100 µg PM | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 18/23 | 18/24 | 16/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 µg AM (N=23) | FF 100 µg PM (N=24) | Placebo (N=25)
Viral upper respiratory tract infection (Infections and infestations) | 1 | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0
Headache (Nervous system disorders) | 12 | 10 | 9
Dizziness (Nervous system disorders) | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Oral pruritus (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.